CLINICAL TRIAL: NCT05699434
Title: Obstetrics and Gynecology Residents and Experts' Knowledge of, Attitudes Toward, Practice Behaviors, and Self-confidence Levels of Caring for Lesbian, Bisexual, and Transgender (LBT+) Patients in Turkey; A Descriptive-cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Arnavutkoy EAH
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: LGBT; attitude; knowledge; practice behaviour; self confidence
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstetrics and Gynecology residenst and experts: Obstetrics and Gynecology residents and expert knowledge of, attitudes toward, practice behaviors, and self-confidence levels of caring for lesbian, bisexual, and transgender (LBT+) patients in Turkey ( Istanbul)
  Interventions: Behavioral: Obstetrics and Gynecology residents and experts'

INTERVENTIONS:
Behavioral: Obstetrics and Gynecology residents and experts' — Obstetrics and Gynecology residents and experts' knowledge of, attitudes toward, practice behaviors, and self-confidence levels of caring for lesbian, bisexual, and transgender (LBT+) patients in Turkey (Istanbul)

SUMMARY:
Obstetrics and Gynecology residents and experts' knowledge of, attitudes toward, practice behaviors, and self-confidence levels of caring for lesbian, bisexual, and transgender (LBT+) patients in Turkey; A descriptive-cross sectional study

DETAILED DESCRIPTION:
There are various studies about LGBT people's problems while utilizing healthcare services and interactions with physicians in Turkey and other countries. There is a lack in the curriculum for obstetricians and gynecologists regarding LGBT individuals' healthcare problems. In this study, we tried to evaluate obstetrics and gynecology residents/experts' knowledge level about LGBT individuals, attitudes toward these sexual minority individuals in their clinical practices, practice behaviors and experience levels about this condition, and their confidence level about caring for sexual minority individuals by performing cross-sectional study using online survey platform.

ELIGIBILITY:
Inclusion Criteria:

* work actively as an Obstetrician and Gynecologist in Istanbul/Turkey

Exclusion Criteria:

* retired clinicians
* LGBT individuals working as Obstetrician and Gynecologist

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Turkish Obstetrics and Gynecologists (residents and experts) working active in Istanbul
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Obstetrics and Gynecology residents and experts' knowledge of, attitudes toward, practice behaviors, and self-confidence levels of caring for lesbian, bisexual, and transgender (LBT+) patients | Time Frame: 2 months
  self produced questionnares evaluating Obstetricians and Gynecologists knowledge,self confidence,practice behaviour and attitude toward LGBT individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No